CLINICAL TRIAL: NCT06093919
Title: Study of Prevalence of Eating Disorder in Liver Transplant Patients
Acronym: Pré-THETA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Other Study IDs: F20230719110020
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Eating Disorders; Eating Disorder Binge; Liver Transplant; Complications; Alcohol Use Disorder; Cirrhosis Alcoholic
MeSH Terms: conditions — Feeding and Eating Disorders; Binge-Eating Disorder; Alcoholism; Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant patients: This cohort will consist of all liver transplant patients followed between 01/01/2023 and 06/30/2024

SUMMARY:
The main goal of this observational study is to measure the prevalence of binge eating disorder in liver transplant patients by evaluating the responses to the Bulimia Test.

Secondary objectives of the study are to:

* Determine the prevalence of binge eating disorders in liver transplant patients following alcoholic cirrhosis, evaluated by the Bulimia Test;
* Study the association between the presence of eating disorder behaviours and liver damage : hepatic steatosis and fibrosis determined by Fibroscan (Transient elastography and controlled attenuation parameter)
* Study the association between presence of eating disorder behaviours and alcohol use disorder, measured by Alcohol Use Disorders Identification Test-Consumption

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* had a liver transplant and followed at University Hospital of Poitiers
* responded to the Bulimia Test-Revised and to the Alcohol Use Disorders Identification Test-Consumption
* had a Fibroscan within the year

Exclusion Criteria:

* Patient without Fibroscan and not responded to both scale : Bulimia Test-Revised and Alcohol Use Disorders Identification Test-Consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all liver transplant patients at the University Hospital of Poitiers followed between 01/01/2023 and 06/30/2024
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of binge eating disorder in liver transplant patients | 1 year
  The prevalence is defined as the percentage of liver transplant patients with a score higher than 88 on the Bulimia Test-Revised. The Bulimia Test-Revised is a validated test. It is a 36 item self-report questionnaire to assess the presence of bulimic symptoms. Scores range from 29-140 with those greater than 104 being indicative of bulimia nervosa.

SECONDARY OUTCOMES:
Prevalence for binge eating disorder in liver transplant patients following alcoholic cirrhosis | 1 year
  The prevalence was defined as the percentage of liver transplant patients following alcoholic cirrhosis with a score higher than 88 on the Bulimia Test-Revised. The Bulimia Test-Revised is a validated test. It is a 36 item self-report questionnaire to assess the presence of bulimic symptoms. Scores range from 29-140 with those greater than 104 being indicative of bulimia nervosa.
Correlation between the BulimiaTest-Revised score and liver damage determined by the Fibroscan | 1 year
  The Correlation was defined by the coefficient between the bulimia-Test score and the liver damage defined by the levels of hepatic steatosis and fibrosis witch are measured by Transient elastography and controlled attenuation parameter using Fibroscan. The Bulimia Test-Revised is a validated, it is a 36 item self-report questionnaire to assess the presence of bulimic symptoms. Scores range from 29-140 with those greater than 104 being indicative of bulimia nervosa.
Correlation between the Bulimia-Test score and the Alcohol Use Disorders Identification Test-Consumption score | 1 year
  The Correlation was defined by the coefficient between the bulimia-Test score and the Alcohol Use Disorders Identification Test-Consumption score. The Bulimia Test-Revised is a validated. It is a 36 item self-report questionnaire to assess the presence of bulimic symptoms. Scores range from 29-140 with those greater than 104 being indicative of bulimia nervosa.
  The Alcohol Use Disorders Identification Test-Consumption score is a validated test. It's scored on a scale of 0-12 (scores of 0 reflect no alcohol use). For men, a score of 4 or more is considered positive; for women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely the patient's drinking is affecting his/her health and safety.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Henri Laborit, Poitiers
  - University Hospital of Poitiers (CHU de Poitiers), Poitiers

IPD SHARING:
Plan to Share IPD: Undecided